CLINICAL TRIAL: NCT03071419
Title: Father-Focused Nutrition and Parenting Program to Help Prevent Childhood Obesity in Preschool Age Children
Brief Title: A Nutrition and Parenting Program for Fathers and Their Pre-school Age Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amy Mobley, Assistant Professor, University of Connecticut
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H15-338; 1R21HD087817-01 (NIH)
Record Dates: First submitted 2017-02-26; First posted 2017-03-06 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Pediatric Obesity
Keywords: fathers
MeSH Terms: conditions — Pediatric Obesity | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The interventionists will not be aware of whether participants are in the intervention or wait-list control group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutrition and Parenting Intervention (Experimental): Participants (n=30, father/child dyads in groups of 10) will receive an 8 session (2 hours/session) community-based intervention including nutrition and parent education with between-session technology enhancements.
  Interventions: Behavioral: Nutrition and Parenting Intervention
- Wait-list Control (Active Comparator): Participants (n=30, father/child dyads in groups of 10) will serve as a wait-list control group and receive the same Nutrition and Parenting Intervention after completing pre and post assessments several weeks apart.
  Interventions: Behavioral: Nutrition and Parenting Intervention

INTERVENTIONS:
Behavioral: Nutrition and Parenting Intervention — The proposed intervention will evaluate and explore the unique influences that low-income fathers have on their preschool age children's obesogenic behaviors and obesity risk.

SUMMARY:
This pilot study evaluates the feasibility and impact of a father-focused childhood obesity prevention program on paternal food-related parenting practices, mealtime behaviors and father/child nutrition and physical activity behaviors. Half of participants (low-income father and child dyads) will receive an intervention immediately while the other half of participants will serve as a wait-list control group and receive the intervention at a later date.

DETAILED DESCRIPTION:
All participants (low-income father and child dyads) will receive an 8 session (2 hours/session) (DAD) including community-based, hands-on, nutrition and parent education intervention with between-session technology enhancements. Dyads will be randomly assigned within groups of 10 to DAD or a wait-list control group (DELAY). Assessments will be conducted at pre, post and 1 month post including a subset of data from cohabiting mothers to assess moderating influences on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* "Father" eligible for a federal food assistance or related program (e.g. SNAP) or living in an area with >30% poverty
* Having at least one preschool age child (ages 3-5 years old)
* At least 18 years of age and able to speak English

Exclusion Criteria:

* No presence or interaction with child during meal or snack times.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — "Father" will be defined as the main male figure with a relationship with the preschool aged child. This includes biological fathers, live-in boyfriends, stepfathers, grandfathers or other father figures.
Enrollment: 72 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Comprehensive Feeding Practices Questionnaire | Change from baseline at 8 weeks
  Food-related parenting practices including parental support, control, structure, feeding

SECONDARY OUTCOMES:
Father & child diet quality | Change from baseline at 8 weeks
  Diet quality assessed using Healthy Eating Index (24 hour recall)
Father & child BMI/BMI Z-Score | Change from baseline at 8 weeks
Meals in Our Household questionnaire | Change from baseline at 8 weeks
  Mealtime behaviors and practices including shopping, meal planning, cooking, family meals
Healthy Kids Questionnaire | Change from baseline at 8 weeks
  Father and child nutrition behaviors including vegetable and sweetened beverage intake frequency & Physical activity behaviors including play and screen time

CONTACTS AND LOCATIONS:
Overall Officials: Amy R Mobley, PhD, RD, Principal Investigator — University of Connecticut
Locations (2):
- United States (2):
  - Hockanum School, Head Start Program, East Hartford, Connecticut
  - Manchester Preschool Center, Manchester, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mobley AR, Gans KM, Adamsons K, Huedo-Medina TB. Feasibility, Acceptability, and Preliminary Outcomes of a Father-Focused Childhood Obesity Prevention Program for Low-Income Families with Preschool-Age Children. Child Obes. 2023 Jan;19(1):13-24. doi: 10.1089/chi.2021.0225. Epub 2022 Mar 11. PMID 35275734